CLINICAL TRIAL: NCT05897528
Title: Impaired Insulin Regulation Determining Severity of Severe Acute Respiratory Syndrome COVID-19 Infection Confounded by Ethnicity
Brief Title: Insulin Regulation and Severity of Severe Acute Respiratory Syndrome COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-35
Record Dates: First submitted 2023-05-24; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; Diabetes Mellitus; COVID-19 Pneumonia; COVID-19 Respiratory Infection
MeSH Terms: conditions — COVID-19; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetes Mellitus Positive Group: All patient that have a diagnosis of diabetes mellitus and COVID-19 Diagnosis
  Interventions: Other: No Intervention
- Diabetes Mellitus Negative Group: All patient that do not have a diagnosis of diabetes mellitus but do have a diagnosis of COVID-19.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Difference in outcomes in patients with COVID-19 diagnosis and diabetes mellitus groups

SUMMARY:
The Coronavirus Disease of 2019 (COVID-19) pandemic has caused an international healthcare crisis and produced a large healthcare burden. Diabetes mellitus is a common disease that can be controlled via pharmacologic agents; however, many patients have poor glycemic control, leading to disease-related complications. Diabetes mellitus has been reported in the literature to be associated with increasing morbidity and mortality in COVID-19 patients, and some hypothesize that this is due to insulin dysregulation propagating a pro-inflammatory state. The investigators aim to contribute to the growing body of literature that assesses the associations between glucose homeostasis and COVID-19 disease severity and mortality.

DETAILED DESCRIPTION:
The Coronavirus Disease of 2019 (COVID-19) is caused by an infection from the severe acute respiratory syndrome coronavirus 2, and the first case in the United States was documented on January 31, 2020. Severe acute respiratory syndrome coronavirus 2 is a RNA virus that has 82% homology with severe acute respiratory syndrome coronavirus 2, which caused a pandemic in 2003. Severe acute respiratory syndrome coronavirus 2 enters cells via the angiotensin converting enzyme 2 (ACE2) receptor, which is primarily expressed in the lung. COVID-19 has led to a worldwide pandemic, with over six million deaths attributed to the virus, according to the World Health Organization. This emerging infection has caused an international healthcare crisis with a significant burden on healthcare workers.

Advanced age, male sex, cardiovascular disease, and diabetes mellitus are known to be associated with increasing risk for COVID-19 severity and mortality. Diabetes mellitus is a common disease that affects the general population by disrupting glucose homeostasis. Impaired glycemic control produces a state of hyperglycemia, which leads to multi-organ injury via a chronic, pathophysiologic inflammatory state. Early retrospective studies demonstrated the association of insulin dysregulation with COVID-19 disease severity and mortality. With more data availability and time, many studies have been conducted to better characterize the relationships between hyperglycemia and elevated hemoglobin A1c (HbA1c) with COVID-19 disease susceptibility, severity, and mortality.

Through this retrospective analysis, the investigators investigate the associations of HbA1c levels and hyperglycemia with COVID-19 mortality and disease severity.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* COVID-19 confirmed by laboratory testing (ICD10 U07.1)
* Pneumonia due to COVID-19 (ICD10 J12.82)
* Diagnosis of Diabetes Mellitus

Exclusion Criteria:

* All patients under the age of 18
* COVID in pregnancy

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: To evaluate diabetes mellitus and the associations with COVID-19 disease severity in patients older than 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Total time frame was 360 days
  The time spent hospitalized in days.
Length of time spent intubated on a ventilator | 30 days
  The time spent intubated on a ventilator in days.
Hospital Mortality | 30 days
  Survival within the first 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Phan, MD, Principal Investigator — Arrowhead Regional Medical Center
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar A, Arora A, Sharma P, Anikhindi SA, Bansal N, Singla V, Khare S, Srivastava A. Is diabetes mellitus associated with mortality and severity of COVID-19? A meta-analysis. Diabetes Metab Syndr. 2020 Jul-Aug;14(4):535-545. doi: 10.1016/j.dsx.2020.04.044. Epub 2020 May 6. PMID 32408118
- [Background] Espinosa OA, Zanetti ADS, Antunes EF, Longhi FG, Matos TA, Battaglini PF. Prevalence of comorbidities in patients and mortality cases affected by SARS-CoV2: a systematic review and meta-analysis. Rev Inst Med Trop Sao Paulo. 2020 Jun 22;62:e43. doi: 10.1590/S1678-9946202062043. eCollection 2020. PMID 32578683
- [Background] Fox T, Ruddiman K, Lo KB, Peterson E, DeJoy R 3rd, Salacup G, Pelayo J, Bhargav R, Gul F, Albano J, Azmaiparashvili Z, Anastasopoulou C, Patarroyo-Aponte G. The relationship between diabetes and clinical outcomes in COVID-19: a single-center retrospective analysis. Acta Diabetol. 2021 Jan;58(1):33-38. doi: 10.1007/s00592-020-01592-8. Epub 2020 Aug 17. PMID 32804317
- [Background] Apicella M, Campopiano MC, Mantuano M, Mazoni L, Coppelli A, Del Prato S. COVID-19 in people with diabetes: understanding the reasons for worse outcomes. Lancet Diabetes Endocrinol. 2020 Sep;8(9):782-792. doi: 10.1016/S2213-8587(20)30238-2. Epub 2020 Jul 17. PMID 32687793